CLINICAL TRIAL: NCT06615063
Title: Limb Splinting for Intravenous Cannulae in Neonates and Its Effects on Life Span of Intravenous Cannulae; A Randomised Controlled Trial.
Brief Title: Limb Splinting for Intravenous Cannulae in Neonates and Its Effects on Life Span of Intravenous Cannulae
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rawalpindi Medical College (Other)
Responsible Party: Principal Investigator, Hasnain Aslam, Principal Investigator, Rawalpindi Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RMU-RRF-SUR-007-23
Record Dates: First submitted 2024-08-14; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Neonatal Peripheral Intravenous Cannulation; Limb Splinting; Intravenous Cannula Lifespan; Extravasation; Extravasation Injury
Keywords: Neonatal Care; Intravenous Cannulation; Splinting; Neonatal Surgery; Pediatric Surgery; Extravasation

STUDY DESIGN:
Intervention Model Description: The interventional study model of the above article is a Parallel Assignment model.
  In this study, neonates are randomly assigned to one of two groups: one group receives the intervention (limb splinting) while the other group does not (non-splinted). The outcomes (e.g., lifespan of the IV cannula, incidence of complications) are then compared between these two parallel groups to determine the effectiveness of the intervention.
Masking Description: The description of the study does not explicitly mention any masking (blinding).
  In the context provided, the primary investigator collects and analyzes the data using self-designed questionnaires. Typically, in such studies, the intervention (splinting) would be known to the participants and the healthcare providers administering the IV cannulation. Therefore, masking of the participants and providers might not be feasible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Splint Group (Experimental): These neonates receive peripheral intravenous cannulation with limb splinting.
  Interventions: Other: Hasi's Splint
- Non-Splint Group (No Intervention): These neonates receive peripheral intravenous cannulation without limb splinting.

INTERVENTIONS:
Other: Hasi's Splint — A splint made up of cotton and gauze piece rolled over a hard cardboard piece and covered by adhesive tape was applied to the limb immediately after fixing the cannula, as per the standardised method, to prevent movement at the underlying joint. Dimensions of the splints used were standardised as length extending two and a half inches on either side of the joint and width equal to the width of the limb just proximal to the joint.
  Arms: Splint Group

SUMMARY:
The goal of this randomized controlled trial is to assess the effectiveness of limb splinting in increasing the lifespan of intravenous (IV) cannulae in neonates. The study involves neonatal patients requiring peripheral IV cannulation. The main questions it aims to answer are:

Does limb splinting increase the lifespan of IV cannulae compared to non-splinting? What are the effects of splinting on the incidence of complications like extravasation, occlusion, and leakage? Researchers will compare neonates with IV cannulae in splinted limbs to those with IV cannulae in non-splinted limbs to see if splinting extends the cannula's lifespan and reduces complications.

Participants will:

Undergo peripheral IV cannulation with and without limb splinting. Have the lifespan of their IV cannulae monitored and recorded until removal due to various complications or routine changes.

DETAILED DESCRIPTION:
This randomized controlled trial aims to investigate the impact of limb splinting on the lifespan of intravenous (IV) cannulae in neonates. The study is motivated by the need to enhance the efficacy and safety of peripheral IV cannulation in neonates, who frequently require intravenous access for the administration of medications and fluids during hospitalization. Peripheral IV cannulation, although common, is associated with a limited dwell time and various complications, including extravasation, occlusion, and leakage, which can lead to multiple cannulations and increased discomfort for neonates.

The study is designed to compare the lifespan of IV cannulae in neonates who have their limbs splinted with those who do not. The primary focus is on whether splinting the limb can effectively increase the dwell time of the IV cannula, thereby reducing the frequency of cannulation and associated complications. The trial involves 246 neonates, randomly assigned to either the splint or non-splint group, with an equal number of participants in each group.

Neonates included in the study will undergo standard peripheral IV cannulation procedures, with all cannulae being inserted by experienced medical staff under controlled conditions. In the splint group, the limb with the IV cannula will be immobilized using a splint, while in the non-splint group, the limb will not be splinted. The time from cannula insertion to removal will be meticulously recorded for each neonate, along with any complications that arise, such as extravasation, accidental dislodgment, infiltration, phlebitis, leakage, or occlusion.

Data will be collected using a self-designed questionnaire, ensuring that the information is only accessible to the primary investigator to maintain data integrity and confidentiality. The study will employ rigorous statistical analysis, including two-sample t-tests to compare the mean dwell times between the splinted and non-splinted groups, and Spearman's rank analysis to explore correlations between various parameters.

The outcomes of this trial are expected to provide valuable insights into the effectiveness of limb splinting as a technique for increasing the lifespan of IV cannulae in neonates. The findings could potentially influence clinical practices by identifying a simple yet effective method to enhance the safety and comfort of neonatal patients requiring IV therapy.

ELIGIBILITY:
Inclusion Criteria:

* All neonates with intravenous cannulae

Exclusion Criteria:

* All neonates in neonatal ICU
* All neonates with central venous line in place
* All neonates that are on ventilatory support

Ages: 1 Hour to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 246 (Actual)
Dates: Start 2022-12-10 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
lifespan (dwell time) of the intravenous (IV) cannulae. | from 0 to 48 hours
  The study aims to compare the mean dwell time of IV cannulae between the splinted and non-splinted groups to determine if limb splinting has a significant effect on extending the duration for which the cannula remains functional before removal.

SECONDARY OUTCOMES:
Incidence of Complications | from 0 to 48 hours
  Various complications related to IV cannulation are assessed, including:
  Extravasation Accidental Dislodgment Infiltration Phlebitis Leakage Occlusion

CONTACTS AND LOCATIONS:
Overall Officials: Ali Raza Chaudhry, MBBS, MS, Study Director — Rawalpindi Medical College; Mudassar Fiaz Gondal, MBBS, MS, Study Chair — Rawalpindi Medical College; hasnain Aslam, MBBS, Principal Investigator — Rawalpindi Medical College
Locations (1):
- Department of Pediatric Surgery,Holy Family Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Barker DP, Rutter N. Exposure to invasive procedures in neonatal intensive care unit admissions. Arch Dis Child Fetal Neonatal Ed. 1995 Jan;72(1):F47-8. doi: 10.1136/fn.72.1.f47. PMID 7743285
- [Result] Bakr AF. Intravenous lines-related sepsis in newborn babies admitted to NICU in a developing country. J Trop Pediatr. 2003 Oct;49(5):295-7. doi: 10.1093/tropej/49.5.295. PMID 14604163
- [Result] Gupta P, Rai R, Basu S, Faridi MM. Life span of peripheral intravenous cannula in a neonatal intensive care unit of a developing country. J Pediatr Nurs. 2003 Aug;18(4):287-92. doi: 10.1016/s0882-5963(03)00052-6. PMID 12923741
- [Result] Mewahegn AA, Tadesse B, GebreEyesus FA, Tarekegn TT, Amlak BT, Emeria MS, Temere BC, Terefe TF, Zewudie BT, Geletie HA, Mengist ST. Lifespan and Associated Factors of Peripheral Intravenous Cannula Among Hospitalized Children in Public Hospitals of the Gurage Zone, Ethiopia, 2021. Pediatric Health Med Ther. 2022 Mar 25;13:81-93. doi: 10.2147/PHMT.S351759. eCollection 2022. PMID 35368745
- [Result] Franck LS, Hummel D, Connell K, Quinn D, Montgomery J. The safety and efficacy of peripheral intravenous catheters in ill neonates. Neonatal Netw. 2001 Aug;20(5):33-8. doi: 10.1891/0730-0832.20.5.33. PMID 12144220
- [Result] Birhane E, Kidanu K, Kassa M, Gerezgiher D, Tsegay L, Weldu B, Kidane G, Gerensea H. Lifespan and associated factors of peripheral intravenous Cannula among infants admitted in public hospitals of Mekelle City, Tigray, Ethiopia, 2016. BMC Nurs. 2017 Jun 15;16:33. doi: 10.1186/s12912-017-0227-1. eCollection 2017. PMID 28638278
- [Result] Dalal SS, Chawla D, Singh J, Agarwal RK, Deorari AK, Paul VK. Limb splinting for intravenous cannulae in neonates: a randomised controlled trial. Arch Dis Child Fetal Neonatal Ed. 2009 Nov;94(6):F394-6. doi: 10.1136/adc.2008.147595. Epub 2009 May 12. PMID 19439433
- [Result] Morris W, Heong Tay M. Strategies for preventing peripheral intravenous cannula infection. Br J Nurs. 2008 Oct 23-Nov 12;17(19):S14-21. doi: 10.12968/bjon.2008.17.Sup8.31470. PMID 18974681
- [Result] Johnson RV, Donn SM. Life span of intravenous cannulas in a neonatal intensive care unit. Am J Dis Child. 1988 Sep;142(9):968-71. doi: 10.1001/archpedi.1988.02150090066024. PMID 3414629
- [Result] Shenoy S, Karunakar BP. Factors influencing the peripheral venous catheter survival in critically ill children in a pediatric intensive care unit. Indian J Pediatr. 2014 Dec;81(12):1293-6. doi: 10.1007/s12098-014-1430-7. Epub 2014 May 6. PMID 24796410
- [Result] Serane V T, Rajasekaran R, Vijayadevagaran V, Kothendaraman B. Peripheral intravenous cannulae in neonates: To splint or not? J Vasc Access. 2022 May;23(3):398-402. doi: 10.1177/1129729821996926. Epub 2021 Feb 23. PMID 33619983